CLINICAL TRIAL: NCT06339372
Title: Perioperative Supplementation With Immunonutrition and Its Impact on Surgical Outcome and Pain in Oral Cavity or Mandibular Tumours
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Samar Saed Ramadan, Assistant Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Cairo University, Cairo , Egypt., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AP1912-30102
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Immunonutrition; Surgical Outcome; Pain; Oral Cavity; Mandibular Tumor
MeSH Terms: conditions — Pain; Mandibular Neoplasms | interventions — Docosahexaenoic Acids; alanylglutamine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (standard feeding) (Other): Patients received only standard feeding with caloric distribution (45%-50% carbohydrates,20-35% from fats and 10-35% from protein)
  Interventions: Dietary Supplement: Standard feeding
- Group B (immunonutrition mixture) (Experimental): Patients received perioperative supplementation with omega 3 and dipeptiven (immunonutrition mixture) plus standard feeding.
  Interventions: Dietary Supplement: Omega 3 and dipeptiven

INTERVENTIONS:
Dietary Supplement: Standard feeding — Patients received only standard feeding with caloric distribution (45%-50% carbohydrates,20_35% from fats and 10-35% from protein)
  Arms: Group A (standard feeding)
Dietary Supplement: Omega 3 and dipeptiven — Patients received perioperative supplementation with omega 3 and dipeptiven (immunonutrition mixture) plus standard feeding.
  Arms: Group B (immunonutrition mixture)

SUMMARY:
The aim of this study was to investigate the effect of adding omega 3 and dipeptiven to standard feeding in head and neck patients who will undergo oral cavity tumour resection or mandibular tumour resection (immunonutrrition mixture) on wound infection, fistula formation and length of hospital stay ,total dose of intraoperative and postoperative opioids (opioid consumption and pain incidence ,mortality and other postoperative complications as urinary tract infection (UTI) and pneumonia.

DETAILED DESCRIPTION:
Enhanced Recovery after Surgery (ERAS). A series of components that combine to minimize stress and to facilitate the return of function have been described: these include preoperative preparation and medication, fluid balance, anesthesia and postoperative analgesia, pre- and postoperative nutrition, and mobilization.

Nutrition therapy is the provision of nutrition or nutrients either orally (regular diet, therapeutic diet, e.g. fortified food, oral nutritional supplements) or via enteral nutrition (EN) or parenteral nutrition (PN) to prevent or treat malnutrition.

Head and neck cancer surgery usually means surgery to treat cancer of the mouth, throat or larynx . The surgery is complicated and people often experience problems such as wound infections and wound breakdown, as well as infections such as pneumonia.

The use of a nutritional supplement enriched with Omega 3 fatty acids is associated with a greater preoperative weight loss, reduced postoperative pain and decreased postoperative levels of C reactive protein in patients undergoing Roux-en-Y gastric bypass.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years.
* Both sexes.
* American Society of Anesthesiologists (ASA) physical status I or II .
* Patient undergoing mandibular or oral cavity tumour resection.
* Body mass index (BMI) between 18.5-24.9.
* Patient with serum albumen above 3 gm.
* Patient with written valid consent

Exclusion Criteria:

* Patient refusal and uncooperative patients.
* Patient ASA III or IV.
* Age more than 60 or less than 18.
* Serum albumen less than 3.
* Pre-existing severe malnourishment.
* Allergy to test drugs.
* Patients on tranquilizers, hypnotics, sedatives and other psychotropic patient on steroids and NSAID.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 176 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
The incidence of wound infection | 28 days after intervention
  Evidence of redness and tenderness of surgical wound with discharge of pus was defined as a wound infection.

SECONDARY OUTCOMES:
Fistula formation | 28 days after intervention
  Fistula formation was measured postoperatively.
Length of hospital stay | 28 days after intervention
  Length of hospital stay was measured from admission discharge from hospital
Total dose of intraoperative opioids | Intraoperative
  Total dose of intraoperative opioids was calculated in either group
Total dose of postoperative opioids | 12 hours postoperative
  Total dose of postoperative opioids was calculated in either group
Degree of pain | 12 hours postoperative
  Postoperative pain will be assessed by visual analogue scale (VAS) every 4 h. for 12 h. Patients reporting VAS score (more than 3) will receive rescue analgesics. VAS (0 represents "no pain" while 10 represents "the worst pain imaginable").
The incidence of mortality | 28 days after intervention
  Mortality was measured postoperatively
The incidence of complications | 12 hours postoperative
  Postoperative complications as urinary tract infection (UTI)and pneumonia.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author